CLINICAL TRIAL: NCT02961010
Title: A Cluster Randomised Controlled Trial of Keeping Safe: Investigating the Effectiveness of a Whole School Preventative Education Programme in Improving Children's Knowledge and Understanding to Keep Safe in Situations of Abuse
Brief Title: Evaluating the Effectiveness of Keeping Safe - a School Based Intervention Aimed at Preventing Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Society for the Prevention of Cruelty to Children (Other)
Collaborators: Department of Education Northern Ireland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIKS001
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Child Maltreatment
Keywords: school based prevention, child sexual and domestic abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive the Keeping Safe programme between 2016 and 2018. This comprises a blended package of continuing professional development training and support (plus resource materials) for teachers and school staff to enable them teach sensitive preventative education concepts through the formal statutory Personal Development curriculum, and all other informal opportunities that present in the daily life of the school. Following randomisation, intervention schools will receive the package of training and support across a 3 month period and will then implement/teach in their school across 2 school years. The intervention group will collect outcome data for the evaluation between March 2016 and June 2018.
  Interventions: Behavioral: Keeping Safe
- Wait-list Control Group (No Intervention): The Wait List Control group will continue with standard practice of teaching the statutory Personal Development curriculum between 2016 and 2018. They will not receive the Keeping Safe intervention until Sept 2018 following completion of the evaluation. The Waitlist control intervention group will collect outcome data for the evaluation between March 2016 and June 2018.

INTERVENTIONS:
Behavioral: Keeping Safe — A whole school Preventative Education programme
  Arms: Intervention Group

SUMMARY:
This study evaluates the effectiveness of Keeping Safe, a whole school preventative education intervention in improving children's knowledge and understanding to keep safe in situations of abuse. The intervention

* Comprises three themes (1) Healthy Relationships; (2) My Body; and (3) Being Safe and includes content across the following keeping safe concepts; bullying, neglect, emotional, physical, domestic and sexual abuse, in online and offline contexts.
* Includes activities for the formal and informal school curricula - 63 lessons will be taught to children by their classroom teacher; 3 per term, 9 per year across 7 years from Primary 1 to primary 7 (age 4-11 years).
* Each lesson is accompanied by directed homework activities to involve and engage parents and enable them reinforce learning at home. A number of whole school, key stage and year group assemblies have also been prepared.
* At the beginning of each term school leaders will deliver a prepared assembly to introduce the theme for the term. Following this assembly each teacher will deliver 3 lessons tailored to the age group of their class and parents will assist with home works. The lessons use eBooks, character animations, stories, rhymes, and interactive whiteboard activities to engage children in their learning.

The intervention adopts a whole-school approach and seeks to build the capacity and skills of teachers and parents as key partners. Teachers will receive a comprehensive package of training, ongoing support and resource materials to equip them with the skills they need to effectively communicate sensitive keeping safe messages. Parents will also receive a package of resources to help them feel confident about communicating sensitive messages to their children.

DETAILED DESCRIPTION:
Exploratory research, funded by the Department of Education and undertaken by the NSPCC in 2008, investigated the need for preventative education that aimed to equip pupils with the skills to recognise and respond appropriately to bullying, child abuse and domestic abuse in primary schools in Northern Ireland. Subsequently, an intervention was designed based on the findings from stakeholder consultations (NSPCC reports, 2011) and existing research in the field of school based prevention.

This study uses a cluster randomised controlled trial (RCT) design to evaluate the effectiveness of Keeping Safe, a whole school preventative education intervention in improving children's knowledge and understanding to keep safe in situations of abuse including sexual and domestic abuse.

Randomisation will take place at school level. Schools will be allocated either to the intervention group or a waitlist control group. Following randomisation, intervention schools will receive the package of training and support across a 3 month period. This comprises a blended package of continuing professional development training and support for teachers and school staff to enable them teach sensitive preventative education concepts through the formal statutory Personal Development curriculum, and all other informal opportunities that present in the daily life of the school. Intervention schools will then implement the Keeping Safe intervention in their school for 2 school years, between 2016 and 2018.

The Wait List Control group will continue with standard practice, teaching the Personal Development curriculum between 2016 and 2018. Both groups will participate in the evaluation between March 2016 and July 2018 and the wait list control group will receive the programme in Sept 2018.

This RCT will collect data at 3 timepoints: Baseline (March/ June 2016), Time One (May -June 2017) and Time Two (May- June 2018). Outcome data on children's knowledge and understanding will be collected at all 3 time points as will data on (1) teacher confidence and teaching practice, (2) parent confidence and practice, (3) school level administrative data (e.g. incidence of disclosure and referral out) and (4) school climate/organizational culture.

Primary outcomes (childrens)

1. If exposure to the Keeping Safe programme:

   1. Impacts/changes children's self-reported knowledge and understanding of the following keeping safe concepts; bullying, neglect, physical, emotional, domestic and sexual abuse and in what ways?
   2. Impacts/changes children's self-reported self-efficacy to keep safe in situations of bullying, neglect, physical, emotional, domestic and sexual abuse and in what ways?
2. If children's self-reported knowledge and understanding in relation to the above keeping safe concepts changes over the 2 year period that the programme is being implemented and in what ways?
3. If changes in children's knowledge and understanding vary for different groups of children, and in what ways?

Secondary Outcomes (teachers and parents)

1. If engagement with the Keeping Safe programme:

   1. Impacts/changes teachers' self-reported knowledge in teaching keeping safe messages and in what ways?
   2. Impacts/changes teachers' self-reported confidence and comfort in their own skills to manage sensitive issues in relation to Keeping Safe in the classroom and in what ways?
2. How school context factors such as size, sector and management type, and professional experience factors (length of teaching service, nature of role in school) impact on teacher knowledge, comfort and confidence in teaching Keeping Safe messages.
3. If the continuing professional development training and resources specifically designed for the Keeping Safe programme impact on teachers' teacher knowledge, comfort and confidence in teaching keeping safe messages.
4. If implementing the Keeping Safe programme leads to change in school ethos/climate, and if this differs across schools and in what ways?
5. If engagement with the Keeping Safe programme (parent resources and directed homework activities):

   1. Impacts/changes parents' self-reported knowledge of and confidence to communicate with their child about keeping safe messages and in what ways?
   2. Impacts/changes parents' self-reported current and future confidence to communicate with their child about keeping safe messages and in what ways?
6. If reported changes in parents' knowledge and confidence vary for different groups of parents and in what ways?
7. How personal (gender) parenting profile (age of children, no of children, relationship to child) and home context (postcode and household income) factors impact on parents' knowledge and confidence in relation to keeping safe messages.
8. How parents' knowledge and confidence change over the 2 year period that the programme is being implemented and in what ways?

Data will be collected from children using a questionnaire designed to assess their knowledge and understanding of a range of keeping safe concepts and their self-reported self-efficacy to keep safe in unsafe situations. The questionnaire is a composite measure comprising existing and adapted standardised measures across a range of keeping safe concepts.

The content and administration of the questionnaire (online and paper versions available) have been tailored to ensure age and developmental appropriateness (a number of different versions will be used with varying age groups).

All classroom teachers will be invited to complete a self-report questionnaire (online or paper versions available) measuring their confidence, comfort and teaching practices with regards the programme. Fidelity data with regard to completion of continuing professional learning will be collated from the analytics function on the e-learning programme. Self-reported fidelity to programme implementation in the classroom will be collated using a fidelity monitoring form.

Information on school context (size, sector, management type) and professional experience (length of teaching service, nature of role in school) will also be collected to identify if these impact on teacher knowledge and confidence in teaching keeping safe messages.

All parents will be invited to complete a self-report questionnaire (online and paper) to assess their knowledge and confidence to talk to their children about sensitive keeping safe messages.

Information will also be collected on parents' personal profile (gender) parenting profile (age of children, no of children, relationship to child) home context (Postcode and household income) to identify if these make a difference to parent knowledge and confidence in communicating with their child(ren) about keeping safe messages

Additional school-level administrative data will be collected on Free School Meals/ newcomer children, level of Social Service engagement with school (referrals out etc) to see if these types of experience impact on teacher knowledge and confidence in teaching keeping safe messages, and to examine any difference between intervention and wait-list control schools.

ELIGIBILITY:
Inclusion Criteria:

(1) children 4-11 years attending mainstream sector primary school in Northern Ireland whose school has accepted the invitation to take part in the RCT and whose parents have provided consent for their participation.

Exclusion Criteria:

1. children attending special sector primary schools in Northern Ireland.
2. children 4-11 years attending mainstream sector primary school in Northern Ireland whose school has not been invited/ rejected the invitation to take part in the RCT
3. children 4-11 years attending mainstream sector primary school in Northern Ireland whose school has accepted the invitation to take part in the RCT and whose parents have not provided consent for their participation.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6300 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Children's Knowledge of Abuse Questionnaire (CKAQ) (Tutty, 1995) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  a 33-item self-report measure used to assess children's knowledge of sexual abuse.
Knowledge/Attitudes to Woman Abuse' sub-scale of the 'Child/Teen Witness to Woman Abuse questionnaire (Sudermann et al., 2000) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  a 10-item sub-scale used to assess children's knowledge of Domestic Abuse
Self-Efficacy Sub-scale (Dake et al., 2003) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  a 5-item sub-scale used to assess children's perceived self-efficacy to keep safe in situations of abuse. An additional 4 items were added to this measure concerning online abuse, cyberbullying, and neglect
The What-If Situations Test (WIST) (Saslawsky & Wurtele, 1986) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  a 6-item scenario-based measure designed to assess children's (aged 5-12) ability to recognise and respond to hypothetical situations of abuse. An additional 5 scenarios concerning non-contact, online, and peer-to-peer abuse
two Global Items from the Olweus (1996) bullying questionnaire | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  used to assess frequency of bullying perpetration/victimization.
Adaptation of the Multidimensional Neglectful Behaviour Scale (Kantor et al., 2004) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  This 38-item measure is used as a screening tool for neglect. This measure has been adapted to be used as knowledge measure. 10 items across a range of neglect concepts will be used and presented as true/false questions.
Administrative school level data on children's behaviour | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  to be collated as a proxy measure of skills in recognising, telling and reporting abusive behaviour. This includes child in need/ child at risk disclosures, concerns raised, support received from external agencies.
Revised Children's Manifest Anxiety Scale (RCMAS 2) short 10 item (Reynold and Paget (1981) | twice across 2 years; time 1 May/June 2017, time 2 May/June 2018
  a 10 item short version of the RCMAS - 'What I Think and Feel' used to assess children's self-reported anxiety

SECONDARY OUTCOMES:
Survey on Perceived Confidence in, and Attitudes towards approaches to Teaching and Learning about Sensitive Issues in Health & Personal Development (Lynagh et al., 2010) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  is 26-item survey designed to assess teachers' confidence in teaching and managing sensitive issues in the Health & Personal Development syllabus. Part 2 of this measure will be used to assess teachers' confidence in managing sensitive issues. It has been adapted to focus on the classroom management issues that pertain to the Keeping Safe intervention
Subscale of the Teacher Willingness to Teach Sexual Health Education Questionnaire (Cohen et al., 2012) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  includes a teacher comfort subscale comprising 26-items. This subscale has been adapted to include topics specific to the Keeping Safe programme.
The School Level Environment Survey (SLEQ) (Rentoul & Fraser, 1983; Aldridge et al., 2006) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  a 24 item measure that assesses school culture from the perspective of the teacher. This will be adapted to ensure it is culturally appropriate.
Teacher fidelity measure | 3 times across 2 years; time 0 November/December 2016, time 1 May/June 2017, time 2 May/June 2018
  to completion of the CPD training programme and implementation /teaching of keeping safe programme
Adaptation of 2 scales from the Parenting and Child Sexuality Questionnaire (Morawska et al., 2015) | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  adapted to include topics specific to the Keeping Safe Programme. This measure will be used to assess parent's knowledge and confidence to talk to their children about sensitive keeping safe issues
Parents' current and future confidence measure (Walsh et al., 2012). | 3 times across 2 years; time 0 baseline March/June 2016, time 1 May/June 2017, time 2 May/June 2018
  2 questions adapted to assess parents' current and future confidence to talk to their children about keeping safe

CONTACTS AND LOCATIONS:
Overall Officials: Aisling M McElearney, PhD, Principal Investigator — National Society for the Prevention of Cruelty to Children
Locations (1):
- National Society for the Prevention fo Cruelty to Children, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dake JA, Price JH, Murnan J. Evaluation of a child abuse prevention curriculum for third-grade students: assessment of knowledge and efficacy expectations. J Sch Health. 2003 Feb;73(2):76-82. doi: 10.1111/j.1746-1561.2003.tb03576.x. PMID 12643023
- [Background] Sudermann M, Marshall L. and Loosely S. Evaluation of the London (Ontario) community group treatment programme for children who have witnessed woman abuse. Journal of Aggression, Maltreatment and Trauma 3(1): 127-146, 2000.
- [Background] Tutty L. The revised Children's Knowledge of Abuse Questionnaire: development of a measure of children's understanding of sexual abuse prevention concepts. Social Work Research 19(2): 112-120, 1995.
- [Background] Lynagh M.Gilligan G. and Handley T. Teaching about, and dealing with, sensitive issues in schools: How confident are pre-service teachers? Asia-Pacific Journal of Health, Sport and Physical Education 1 (3/4) 2010
- [Background] Olweus D. The revised Olweus Bully/Victim Questionnaire for Students. Bergen, Norway: University of Bergen.1996
- [Background] Cohen JN. Byers SE. and Sears HA. Factors Affecting Canadian Teachers' Willingness to Teach Sexual Health Education. Sex Education: Sexuality, Society and Learning, 12 (3): 299-316, 2012.
- [Background] Kantor GK, Holt MK, Mebert CJ, Straus MA, Drach KM, Ricci LR, MacAllum CA, Brown W. Development and preliminary psychometric properties of the multidimensional neglectful behavior scale-child report. Child Maltreat. 2004 Nov;9(4):409-28. doi: 10.1177/1077559504269530. PMID 15538039
- [Background] Aldridge JM. Laugksch RC and Fraser BJ School -level environment and outcomes - based education in South Africa. Learning Environment Research 9: 123-147. 2006
- [Background] Walsh K, Brandon L, Chirio L. Mother-child communication about sexual abuse prevention. J Child Sex Abus. 2012;21(4):399-421. doi: 10.1080/10538712.2012.675424. PMID 22809046
- [Background] Saslawsky DA, Wurtele SK. Educating children about sexual abuse: implications for pediatric intervention and possible prevention. J Pediatr Psychol. 1986 Jun;11(2):235-45. doi: 10.1093/jpepsy/11.2.235. No abstract available. PMID 3723285
- [Background] Morawska A, Walsh A, Grabski M, Fletcher R. Parental confidence and preferences for communicating with their child about sexuality. Sex Education 15(3): 235-48, 2015.
- [Background] McElearney A, Scott J, Adamson G, Turtle K, McBride O, Stephenson P. Keeping safe: establishing the need to teach 'keeping safe' messages in primary schools in Northern Ireland: what do children currently know and understand? London: NSPCC, 2011.
- [Background] Stephenson P, McElearney A, Stead J. The development of effective preventative education in primary schools in Northern Ireland: summary report. London: NSPCC, 2011.
- [Background] McElearney A, Stephenson P, Adamson G. The development of effective preventative education in primary schools in Northern Ireland: exploring practice, policy and research implications. London: NSPCC, 2011.
- [Background] McElearney A, Scott J, Stephenson P, Tracey A, Corry D. The views of principals, teachers and other school staff in relation to teaching "keeping safe" messages in primary schools in Northern Ireland. London: NSPCC, 2011.
- [Background] Stephenson P, Tracey A, McElearney A. The views of cross-sector stakeholders in relation to teaching "keeping safe" messages in primary schools in Northern Ireland. London: NSPCC, 2011.
- [Derived] McElearney A, Brennan-Wilson A, Murphy C, Stephenson P, Bunting B. Cluster randomised controlled trial of 'whole school' child maltreatment prevention programme in primary schools in Northern Ireland: study protocol for Keeping Safe. BMC Public Health. 2018 May 3;18(1):590. doi: 10.1186/s12889-018-5492-8. PMID 29724196
- See also: Click here for more information about this study: Preventative 'Keeping Safe' Education in Northern Ireland — http://www.nspcc.org.uk/keeping-safe-NI
- See also: Department of Education website — https://www.education-ni.gov.uk/articles/preventative-education